CLINICAL TRIAL: NCT00361686
Title: Randomized Double Blind Study Comparing Patient Controlled Analgesia With Tramadol vs. Remifentanyl for Women Undergoing 2nd Trimester Abortions
Brief Title: Comparison of Tramadol vs Remifentanyl Patient Controlled Analgesia for Second Trimester Abortions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3820
Record Dates: First submitted 2006-08-06; First posted 2006-08-08 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2006-07

CONDITIONS: Abortion,Induced
Keywords: tramadol; remifentanyl; patient controlled analgesia; abortion
MeSH Terms: interventions — Tramadol; Remifentanil

INTERVENTIONS:
Drug: tramadol
Drug: remifentanyl
Device: patient contolled analgesia

SUMMARY:
Patients undergoing second trimester abortions will recieve either patient controlled analgesia with either remifentanyl or tramadol for pain alleviation.

We beleive both to be equally effective for pain alleviation.

DETAILED DESCRIPTION:
Women undergoing second trimester abortions will recieve patient controlled analgesia eith either tramadol or remifentanyl.

Patients will not know what they are recieving.

Patients in the tramadol goup will get a loading dose of tramadol and metocloparamide while the women in the remifentanyl group will be given a loading placebo.

Women will then be attached to one of the two patinet controlled analgesia protocols.

Throughout their laboring process they will be monitored for blood pressure, pulse, breathing rate, sedation score and nausea.

Additional medicatyion will be given for nausea.

If woman are still in pain the patient controlled analgesia settings will be set to deliver a higher dose. If the woman remains in pain, she will be given an additional per os medication.If this still does not alleviate pain, the option of epidural analgesia will be offered.

ELIGIBILITY:
Inclusion Criteria:

Woman undergoing 2nd trimester abortion -

Exclusion Criteria:

* Seizure disorder

  - * Psychiatric disorder
* Inability to recieve patient controlled analgesia
* Allergy to tramadol or remifentanyl

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction
VAS scores
Nausea
Sedation

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Orbach-Zinger, Study Director — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petach Tiqvah, Israel